CLINICAL TRIAL: NCT05089214
Title: Diagnostic Efficacy Assessment of Two Oral Telemedicine Tools Compared to Intra Oral Clinical Examination Used as a Reference: a Pilot Study in Region Grand-Est
Brief Title: ONE-1 Oral graNd Est 1
Acronym: ONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr. Céline CLEMENT, Head of Dental Public Health Department, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A01306-35
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Dental Decay; Periodontal Abscess; Periodontitis; Gingivitis; Dental Plaque; Calculus, Dental; Missing Teeth
Keywords: Telemedecine; Dental Camera; Nursing Home; Dental Decay; Oral Status
MeSH Terms: conditions — Dental Caries; Periodontal Abscess; Periodontitis; Gingivitis; Dental Plaque; Dental Calculus; Anodontia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intra oral clinical examination (Experimental)
  Interventions: Device: Intra oral cameras

INTERVENTIONS:
Device: Intra oral cameras — Diagnostic comparison of two intra oral cameras

SUMMARY:
This study is about the assessment of two oral telemedecine tools compared to an intra oral clinical examination used as a reference among elderly persons living in nursing home. Our hyposthesis is that the diagnostic performance of the two devices will be similar.

The main goal of the study is to assess the performances of two intra-oral cameras compared to an intra oral clinical examination to detect at least one decayed tooth.

The secondary objectives of this study are :

At patient's level:

1. To assess the performances of two intra-oral cameras types compared to an intra oral clinical examination for detecting each of the following conditions: (i) at least one filled tooth, (ii) at least one missing tooth, (iii) gingivitis, (iv) an abscess, (v) dental plaque and (vi) calculous
2. To assess the concordance between each intra oral cameras and the intra oral clinical examination in the evaluation of the number (i) of decayed teeth, (ii) filled teeth and (iii) missing tooth
3. From video acquisitions of each intra oral cameras, to assess the inter-observer concordance for the diagnostic of each dental pathologies (presence of at least one decayed tooth, filled or missing) and periodontal (presence of gingivitis, abscess, dental plaque or scale)
4. From video acquisitions of each intra oral cameras, to assess the inter-observer agreement of the number of teeth: (i) decayed, (ii) filled and (ii) missing

   At tooth level :
5. To assess the performances of two intra-oral cameras types compared to an intra oral clinical examination for detecting each of the following conditions: (i) a cavity, (ii) a filled tooth and (iii) missing tooth

   In all patients :
6. To assess patient's feelings about the use of each intra oral cameras
7. To compare the time required for video acquisitions between each of intra oral cameras

For patients with dental or periodontal pathologies observed during the intra oral examination:

8 To assess, 2 months after initial evaluation, the proportion of patients attended dental or periodontal care and for which an appointment with a dentist has been scheduled

ELIGIBILITY:
Inclusion Criteria:

* Be an adult person
* Be affiliated of granted of health insurance
* Be resident of a nursing home
* People (or the guardian) who received complete information about the research and who signed the consent form.

Exclusion Criteria:

* People deprived of their liberty by justice's decision, or people following psychiatric treatment according to articles L. 3212-1 et L. 3213-1 of the French law
* People with insufficient skills in French
* People with total bimaxillary prosthesis
* People without any teeth

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Detection of at least one decayed tooth in the mouth of each elderly of the study | within 2 weeks
  * During the intra-oral examination (reference investigation)
  * Using video records of first camera told Soprocare®
  * Using video records of second camea told "wide public"

SECONDARY OUTCOMES:
Conditions of the elderlies of the study will be evaluated thanks to the intra oral clinical examination and the video records of each of the two cameras. | within 2 weeks
  The presence of at least one filled tooth, the absence of at least one tooth, the presence of gingivitis, of an abscess, of dental plaque and calculous in the elderlies of the study will be evaluated thanks to the intra oral clinical examination and the video records of each of the two cameras.
The number of decayed, filled, missing teeth in the elderly of the study will be recorded thanks to the intra oral clinical examination and the video records of each of the two cameras. | within 2 weeks
Presence of each dental conditions (at least one tooth decayed, filled, missing) and each periodontal conditions will be assess by to independent reviewers from video records of each camera. | within 2 weeks
  periodontal conditions = presence of gingigivitis, abscess, dental plaque or calculous
Number of teeth showing each dental conditions (at least one tooth decayed, filled, missing) will be assess by two independent reviewers from video records of each camera. | within 2 weeks
Presence of a decayed, a filled, or missing tooth, will be assess for each tooth of elderly of the study during the clinical examination and the records of each camera. | within 2 weeks
Feeling of the patient will be evaluated thanks to a questionnaire "questionnaire of acceptability of patient's examination" | within 2 weeks
  Each examination (e.g clinical exam, camera 1, camera 2) are evaluated by 8 questions rated from 1 to 6, i.e a score between 8 to 48 for each exam. The questionnaire is an adaptation of the "Whole Systems Demonstrator Service User Technology Acceptability" questionnaire from Hirani, S. P., Rixon, L., Beynon, M., Cartwright, M., Cleanthous, S., Selva, A., Sanders, C. and Newman, S. P. (2016). Quantifying beliefs regarding telehealth: Development of the Whole Systems Demonstrator Service User Technology Acceptability Questionnaire. Journal of Telemedicine and Telecare, 23(4), pp. 460-469. doi:
  10.1177/1357633X16649531
Number of decayed, filled, missing teeth in the elderly of the study will be recorded thanks to the intra oral clinical examination and the video records of each of the two cameras. | within 2 weeks
Number of appointment programation | within 2 weeks
  If a dental or periodontal condition has been brought to light during the intraoral clinical examination, the coordinating physician will assess by phone if the needed care have been realized during the two-month following this examination. If hasn't been realized during this two-month follow-up time, coordinating physician will record if an appointment has been programmed for this needed care.

CONTACTS AND LOCATIONS:
Locations (1):
- EHPAD St Georges, Hannonville-sous-les-Côtes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Veynachter T, Sural Y, Baudot P, Remen T, Baudet A, Kabuth B, Clement C. Diagnostic performance of two teledentistry tools in elderly care facilities: the ONE-1 protocol for a pilot prospective diagnostic study. BMJ Open. 2023 Apr 3;13(4):e063906. doi: 10.1136/bmjopen-2022-063906. PMID 37012012